CLINICAL TRIAL: NCT05645640
Title: China Patient-centered Evaluative Assessment of Cardiac Events (PEACE): Strategy for Cardiovascular Disease Prevention Through Tailored Health Management and Its Effectiveness Assessment Through a Cluster Randomized Trial in Individuals With Elevated Risk (SMARTER)
Brief Title: Strategy for Cardiovascular Disease Prevention Through Tailored Health Management in Individuals With Elevated Risk
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Xi Li, Vice Director of National Clinical Research Center for Cardiovascular Diseases, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-GSP-GG-4
Record Dates: First submitted 2022-11-23; First posted 2022-12-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Risk Reduction; Primary Prevention
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Subjects in the intervention group will receive village doctor-led tailored health management which includes five main components (marking of individual risk factor profiles, tailored targets for risk factor modification, individualized health education based on Smart Phones, health monitoring and feedback based on Smart Bands, and incentive based on gamification).
  Interventions: Combination Product: Village doctor-led tailored health management
- Control (No Intervention): Subjects in the control group will receive usual care (advice on lifestyle change, medication, and rehabilitation).

INTERVENTIONS:
Combination Product: Village doctor-led tailored health management — Investigators will "sketch" features of cardiovascular risk factor combinations for the high-risk subjects and accordingly set tailored promotion targets for them. Subjects will receive individualized consultation about their cardiovascular risk profile and tailored health management led by village doctors. They will receive tailored health text messages pushed by village doctors 3 times a week, including contents in physical activity, healthy diet, smoking abstinence, responsible alcohol drinking, sleep, and medication adherence. They will be provided with a smart band, and supposed to daily wear the smart band to collect health data. The progress of tailored promotion targets will be evaluated every 3 months, and feedback will be given in the form of virtual rewards and punishments: completed (a virtual golden egg) and failed (a virtual bomb). According to the number of virtual golden eggs, participants could redeem project gift in real life.
  Arms: Intervention

SUMMARY:
The China PEACE SMARTER trial is a cluster ramdomized trial aiming to assess the effectiveness of village doctor-led tailored health management on risk reduction of high-risk individuals for cardiovascular disease.

DETAILED DESCRIPTION:
In this study, investigators aim to develop a series of intervention strategies for cardiovascular disease (CVD) prevention through village doctor-led tailored health management in individuals with elevated risk, then assess their effectiveness through a cluster randomized trial. Investigators hypothesize that the village doctor-led tailored health management can reduce the CVD risk and improve risk factor control of the high-risk subjects through 12 months of follow-up. Around 4200 subjects from 120 villages in mainland China who are considered to be eligible according to inclusion and exclusion criteria will be enrolled to the study. The eligibility criteria is: Individuals aged 35 or above who are in high risk for CVD (10-year ASCVD risk ≥10%), able to use smart phone, and contracted with the local family doctor. Patients with history of CVD or severe illnesses, pregnancy, cognition or communication problems are excluded from the study. The selected villages will be assigned (1:1) to either control group (usual care) or intervention group (village doctor-led tailored health management). The primary outcome is the change in 10-year ASCVD risk from baseline to 12 months. Follow up visits will be conducted every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35 or above;
* High CVD risk which defined as 10-year ASCVD risk ≥10% based on China-PAR prediction model;
* Ownership of a smart phone and being able to use apps;
* Being contracted with the local family doctor (village doctor);
* Willing to participate and able to sign informed consent.

Exclusion Criteria:

* CVD history, including myocardial infarction (MI), stroke, heart failure, severe arrhythmia, or peripheral artery disease, or having received percutaneous coronary intervention (PCI) or coronary artery by-pass grafting operation (CABG);
* Severe illnesses, such as cancer, or severe hepatic and renal dysfunction;
* Women during pregnancy, lactation, or plan to have children in the next year;
* Having problems in cognition or communication, or limited daily activities.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4533 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
10-year ASCVD risk score | 12 months
  Changes in 10-year ASCVD risk score from baseline to 12 months

SECONDARY OUTCOMES:
Lifetime ASCVD risk score | 12 months
  Changes in lifetime ASCVD risk score from baseline to 12 months
Blood pressure | 12 months
  Changes in systolic and diastolic blood pressure from baseline to 12 months
Fasting plasma glucose (FPG) | 12 months
  Changes in fasting plasma glucose (FPG) from baseline to 12 months
Non-HDL cholesterol | 12 months
  Changes in Non-HDL cholesterol from baseline to 12 months
Weight change | 12 months
  Changes in proportion of subjects who are overweight and obesity from baseline to 12 months
Smoke abstinence | 12 months
  Changes in proportion of daily smoking persons from baseline to 12 months
Physical activity | 12 months
  Changes in proportion of subjects with insufficient physical activity (<3000 MET min/wk) from baseline to 12 months

OTHER OUTCOMES:
Exploratory Outcome: Medication adherence | 12 months
  Changes in proportion of subjects who report taking the full dose of prescribed medications ≥6 days per week among all necessary subjects from baseline to 12 months
Exploratory Outcome: MACEs | 12 months
  Major adverse cardiovascular events, including occurrence of death, myocardial infarction, stroke, and cardiovascular hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Xi Li, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang X, Wang S, Zhou X, Tang Y, Xing L, Ma S, Xu Y, Wu C, Cui J, Yang Y, Lin C, Wu Y, Zhang H, Fan L, Xu C, Li X; SMARTER Collaborative Group. A village doctor-led mobile health intervention for cardiovascular risk reduction in rural China: cluster randomised controlled trial. BMJ. 2025 May 27;389:e082765. doi: 10.1136/bmj-2024-082765. PMID 40425261